CLINICAL TRIAL: NCT00868205
Title: The Relationship Between Short- and Mid-term Intake of Coffee on in Vivo Levels of Oxidative Stress Parameters in Healthy Adults.
Brief Title: Coffee and In-vivo Oxidative Stress
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Mondelēz International, Inc. (Industry)
Responsible Party: Principal Investigator, W.J. Pasman, TNO, Zeist, The Netherlands, TNO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P8353
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: oxidative stress; Comet assay; antioxidants

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- low coffee dose (Experimental): 3 cups of coffee daily for 8 weeks
  Interventions: Dietary Supplement: Coffee consumption
- high coffee dose (Experimental): 5 cups of coffee daily for eight weeks
  Interventions: Dietary Supplement: Coffee consumption
- Control (No Intervention): Consumption of water instead of coffee daily for eight weeks

INTERVENTIONS:
Dietary Supplement: Coffee consumption — 3 or 5 cups of coffee daily for eight weeks
  Arms: high coffee dose; low coffee dose

SUMMARY:
Food and beverage intake that leads to a decrease in the level of in vivo markers of oxidative stress indicates that such foods and beverages act as antioxidants (AOX) in humans. Coffee drinking at a high level (> 900 ml/day) for a short period of time (1 week) has been shown to reduce DNA oxidative damage-as indicated by a decrease in the level of percent tail DNA (%T)- in study populations comprised mainly of young adults aged < 30 years. It is not clear whether such findings remain present over a longer period of time, and to extend such findings across a population that is more representative of European adults who consume common daily intakes of coffee, which is a low-to-moderate daily intake level (< 750 ml/day). As such, the investigators propose to determine the effect of drinking 3 and 5 cups of coffee per day (equivalent to 450 and 750 ml per day, respectively) for 8-weeks on markers of in vivo oxidative stress relative to control in a population of healthy adults free of chronic diseases aged 35 to 65 years. To ensure that overall health is considered, the investigators will also evaluate the effect on markers of cardiovascular health, inflammation, and glycemic control.

DETAILED DESCRIPTION:
Objective: The main objective of the present study is to determine the short- and mid-term effects of a coffee, on oxidative stress parameters in humans.

Study design: randomized, placebo-controlled, investigator-blinded, 3-arm parallel Study population: 168 apparently healthy volunteers: males and females aged >=35 and <= 65 years.

Intervention: The treatments consist of daily consumption of either:

Treatment 1: 0.45 L coffee (3 cups) and 0.30 L bottled water daily or; Treatment 2: 0.75 L coffee (5 cups) daily or; Treatment 3: 0.75 L water daily Duration of the treatment intervention is 8 weeks. Before the intervention period starts, a run-in period of five weeks where all subjects maintain their low antioxidant diet (Dutch average) is conducted by all subjects in order to standardize the antioxidant intake of the subjects.

Main study parameters/endpoints: Mean level of %T as a measure of DNA oxidative damage at week 8. Secondary outcome is the mean level of 8-isoprostane in 24 hr urine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as assessed by the

   * health and lifestyle questionnaire, (P8353 F02; in Dutch)
   * results of the pre-study laboratory tests
2. Males and females aged >= 35 and <= 65 years at Week 01 of the study
3. Body Mass Index (BMI) >= 20.0 but <= 34.9 kg/m2
4. Blood pressure (automated measurement at site): systolic blood pressure <= 139 mm Hg and diastolic blood pressure <= 89 mm Hg
5. Fasting glucose <= 6.9 mmol/L
6. No smoking or moderate smoking of 1 to 19 cigarettes per day, with the proportion of smokers and nonsmokers representative of the European adult population aged 35-65 years
7. Normal European eating habits as assessed by P8353 F02. Fruit and vegetable consumption at a level representative or less for the European population as assessed by P8353 F06
8. Habitual caffeinated coffee drinker who consumes > 1 cup per day on at least 5 days per week as assessed by P8353 F02
9. Voluntary participation
10. Having given written informed consent
11. Willing to comply with the study procedures
12. Willing to accept use of all nameless data, including publication, and the confidential use and storage of all data for at least 15 years
13. Willing to accept the disclosure of the financial benefit of participation in the study to the authorities concerned.

Exclusion Criteria:

Subjects with one or more of the following characteristics will be excluded from participation:

1. Participation in any clinical trial including blood sampling and/or administration of substances up to 90 days before Day 01 of this study
2. Participation in any non-invasive clinical trial up to 30 days before Day 01 of this study, including no blood sampling and/or oral, intravenous, inhalatory administration of substances
3. Having a history of medical or surgical events that may significantly affect the study outcome (including cardiovascular disease or hypertension at repeated measurements, hypercholesterolemia, hyperglycaemia, kidney or liver disease, cancer, mental illness) based on the health questionnaire
4. Hypertension as indicated by a systolic BP >= 140 mm Hg or a diastolic BP >= 90 mm Hg
5. Hypercholesterolemia as indicated by a fasting LDL-cholesterol >= 4.9 mmol/L at a single screening visit or the use of anti-hypercholesterolemia drugs
6. Diabetes as indicated by a fasting blood glucose >= 7.0 mmol/L at a single screening visit
7. Having (a history of) (severe) gastro-intestinal complaints
8. Using medication for high blood pressure, high cholesterol level, gastro-intestinal complaints, or antidepressants. With the exception of medication for heartburn
9. Not willing to give up the use of coffee, tea, dark chocolate (and foods/beverages containing dark chocolate), vitamin supplements, mineral supplements, herbal products (food, beverage, or supplements), antioxidant dietary supplements, omega-3 fatty acid supplements including flaxseed oil and fish oil supplements, red wine or rose wines, port, sherry, or specific fortified foods
10. Not willing to give up the consumption of coffee beans as food or in foods or the consumption of coffee or espresso in foods (e.g. Tiramisu)
11. The use of any non-study caffeinated/decaffeinated coffee beverage or caffeinated/decaffeinated espresso-based beverage (espresso, cappuccino, latte, frappuccino, or frappe
12. Alcohol consumption > 28 units/week for males and > 21 units/week for females
13. Eating lots of fruit and vegetables (i.e. more than 400 gram vegetables per day and more than 4 servings of fruit per day at screening and during the study. This is twice that of the Dutch dietary recommendations for fruit and vegetable intake)
14. Changing smoking habits (> 5 cigarettes per day)
15. Exercising heavily (> 7 hours/week)
16. Not willing to give up supplement (antioxidant containing) use (to be specified)
17. Reported unexplained weight loss or gain of > 2 kg in the month prior to the pre-study screening
18. Reported slimming or medically prescribed diet
19. Reported vegan, vegetarian or macrobiotic
20. Recent blood donation (<1 month prior to the start of the study)
21. Not willing to give up blood donation during the study.
22. Pregnant or lactating or wishing to become pregnant in the period of the study
23. Personnel of TNO Quality of Life, their partner and their first and second degree relatives
24. Not having a general practitioner
25. Not willing to accept information-transfer concerning participation in the study, or information regarding his/her health, like laboratory results, findings at anamnesis or physical examination and eventual adverse events to and from his general practitioner.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
DNA oxidative damage (Comet assay, %T) | week 0, 4, 5,6,9 and 13

SECONDARY OUTCOMES:
Lipid oxidative damage (8-isoprostane in urine) | week 5,6,9,13

CONTACTS AND LOCATIONS:
Overall Officials: Wilrike Pasman, PhD, Principal Investigator — TNO
Locations (1):
- TNO Quality of Life, Zeist, Utrecht, Netherlands

REFERENCES:
- [Background] Bichler J, Cavin C, Simic T, Chakraborty A, Ferk F, Hoelzl C, Schulte-Hermann R, Kundi M, Haidinger G, Angelis K, Knasmuller S. Coffee consumption protects human lymphocytes against oxidative and 3-amino-1-methyl-5H-pyrido[4,3-b]indole acetate (Trp-P-2) induced DNA-damage: results of an experimental study with human volunteers. Food Chem Toxicol. 2007 Aug;45(8):1428-36. doi: 10.1016/j.fct.2007.02.001. Epub 2007 Feb 12. PMID 17376579
- See also: information about the effect of coffee on antioxidant status — http://www.cosic.org/coffee-and-health/antioxidants